CLINICAL TRIAL: NCT05206734
Title: Incidence of Psychological Comorbidities in Paediatric and Young Adults With Inflammatory Bowel Disease, and the Impacts on Quality-of-life, Disease Severity and Resource Utilisation: A Population-based Cohort Study in the United Kingdom
Brief Title: Risk of Mental Health Conditions in Children and Young Adults With Inflammatory Bowel Disease and Influence on Health
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Optimum Patient Care (Other)
Responsible Party: Sponsor
Other Study IDs: P043
Record Dates: First submitted 2022-01-10; First posted 2022-01-25 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Diseases; Depressive Episode; Recurrent Depressive Disorder; Anxiety Disorder; Psychological Disorder; Self Harm; Suicide, Attempted; Parasuicide; Eating Disorders; Body Image Disorder; Attention Deficit Hyperactivity Disorder; Behavioral Disorder; Adjustment Disorders; Acute Stress Disorder; Schizophrenia; Bipolar Disorder; Post-traumatic Stress Disorder; Sleep Disturbance
MeSH Terms: conditions — Inflammatory Bowel Diseases; Depressive Disorder; Anxiety Disorders; Mental Disorders; Self-Injurious Behavior; Suicide, Attempted; Feeding and Eating Disorders; Body Dysmorphic Disorders; Attention Deficit Disorder with Hyperactivity; Adjustment Disorders; Stress Disorders, Traumatic, Acute; Schizophrenia; Bipolar Disorder; Stress Disorders, Post-Traumatic; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- IBD Cases: All incident cases of Inflammatory Bowel Disease (IBD); comprising of Ulcerative Colitis, Crohn's Disease and IBD Unclassified in children, adolescents and young adults up to their 25th birthday. Cases will be defined based on an algorithm using diagnostic codes from the electronic medical record (EMR).
  Interventions: Other: No specific intervention
- Matched Controls: People without a diagnosis in their electronic medical record (ERM) of Inflammatory Bowel Disease, matched on age group, sex, ethnicity (consistent with UK census categories: White, Asian, Black, Mixed, Other), index of multiple deprivation based on postcode, and by practice where numbers allow.
  Interventions: Other: No specific intervention
- IBD cases with mental health condition: A subset of the IBD cases comprising of those participants with the presence of a mental health condition at the same date as their IBD diagnosis. Mental health defined by the diagnosis of any of depression (recurrent depressive disorder or depressive episode), non-phobia-related anxiety disorder (AD), eating disorders, body image disorder, attention-deficit disorder, behavioural disorders, adjustment disorder, acute stress disorder, schizophrenia, bipolar disorder or post-traumatic stress disorder
  Interventions: Other: No specific intervention
- IBD cases without mental health condition: A subset of the IBD cases comprising of those participants with the absence of a mental health condition at the same date as their IBD diagnosis. Mental health defined by the diagnosis of any of depression (recurrent depressive disorder or depressive episode), non-phobia-related anxiety disorder (AD), eating disorders, body image disorder, attention-deficit disorder, behavioural disorders, adjustment disorder, acute stress disorder, schizophrenia, bipolar disorder or post-traumatic stress disorder
  Interventions: Other: No specific intervention

INTERVENTIONS:
Other: No specific intervention — Observational analysis of usual care only.

SUMMARY:
This study is a large population-based analysis in the United Kingdom (UK) using routine primary care data to investigate the impacts on quality-of-life outcomes and use of healthcare services in people aged 5 - 25 years diagnosed with Inflammatory Bowel Disease (IBD) and the impacts of mental health conditions in those diagnosed with IBD.

DETAILED DESCRIPTION:
This study will use routinely electronic medical record (EMR) data from primary care practices within the Optimum Patient Care Research Database (OPCRD).

Stream 1 primary objective is to compare the prevalence and cumulative incidence of mental health conditions in children, adolescents and young adults (aged 5-25 years) with a diagnosis of Inflammatory Bowel Disease (IBD), compared to matched population controls without a diagnosis of IBD. The secondary objective is to determine the severity of mental health outcomes in those with and without a diagnosis of IBD.

Stream 2 primary objective is to determine the impact of mental health conditions in children, adolescents and young adults (aged 5-25 years) diagnosed with IBD on quality-of-life indicators, such as records for absence from work or school, unemployment, sleep disturbance and substance abuse.

The secondary objectives are to compare indicators of IBD severity, such as medication use, surgical intervention, nutritional supplement prescriptions and markers of nutritional status including underweight or growth retardation,and healthcare resource utilisation.These impacts and indicators will be assessed using participants that have been diagnosed with IBD, comparing those with the presence of a mental health condition to those without a mental health condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 5 years and 25 years
* Registration with a general practices (GP) contributing routinely collected electronic healthcare data to the Optimum Patient Care Research Database (OPCRD) for more than 6 months during the follow up period
* A recorded diagnosis of IBD in the clinical record (cases)

Exclusion Criteria:

• None

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases of IBD in childhood and young adults and age, gender and GP matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 19469 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Principal Investigator — Momentum Data
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
OPCRD data can be access by bone fide researchers for specific research projects subject to approval by Anonymised Data Ethics & Protocol Transparency (ADEPT) Committee. The data used for this study cannot be made available without such approval.
Supporting Information: Study Protocol
Time Frame: The data will be available subject to approval for two years after the study publication date.
Access Criteria: Data sharing is subject to ADEPT Committee approval.

REFERENCES:
- [Derived] Cooney R, Barrett K, Russell RK. Impact of mental health comorbidity in children and young adults with inflammatory bowel disease: a UK population-based cohort study. BMJ Open. 2024 Feb 28;14(2):e080408. doi: 10.1136/bmjopen-2023-080408. PMID 38418244
- [Derived] Cooney R, Tang D, Barrett K, Russell RK. Children and Young Adults With Inflammatory Bowel Disease Have an Increased Incidence and Risk of Developing Mental Health Conditions: A UK Population-Based Cohort Study. Inflamm Bowel Dis. 2024 Aug 1;30(8):1264-1273. doi: 10.1093/ibd/izad169. PMID 37603846

RESULTS

PARTICIPANT FLOW:
Groups:
- Matched Controls: People without a diagnosis in their electronic medical record (ERM) of Inflammatory Bowel Disease, matched on age group, sex, ethnicity (consistent with United Kingdom (UK) census categories: White, Asian, Black, Mixed, Other), index of multiple deprivation based on postcode, and by practice where numbers allow.
  No specific intervention: Observational analysis of usual care only.
Period: Overall Study
Arm/Group | IBD Cases | Matched Controls
Started | 3898 | 15571
IBD Cases With Mental Health Condition | 295 | 0 (Study exposure category: IBD, with or without mental health comorbidity excludes matched controls without IBD)
IBD Cases Without Mental Health Condition | 1648 | 0 (Study exposure category: IBD, with or without mental health comorbidity excludes matched controls without IBD)
Completed | 3898 | 15571
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IBD Cases | Matched Controls | Total
Number analyzed (Participants) | 3898 | 15571 | 19469
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 19 [15 to 21] | 19 [15 to 21] | 19 [15 to 21]
Age, Customized [Count of Participants; unit: Participants]
  Age subgroup: 5-11 years | 364 | 1466 | 1830
  Age subgroup: 12-17 years | 1178 | 4684 | 5862
  Age subgroup: 18-25 years | 2356 | 9421 | 11777
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1819 | 7262 | 9081
  Male | 2079 | 8309 | 10388
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity was categorized to be consistent with the UK official census categories.
  Participants
    Asian or Asian British | 276 | 1000 | 1276
    Black or Black British | 35 | 176 | 211
    White | 1963 | 7536 | 9499
    Mixed | 50 | 136 | 186
    Not stated | 183 | 703 | 886
    Other | 173 | 548 | 721
    Missing | 1218 | 5472 | 6690
Deprivation quintile [Count of Participants; unit: Participants] — Defined using Index of Multiple Deprivation (IMD) derived from the patient's postcode at the point of data extraction.IMD is a measures of relative deprivation.
  Participants
    1 (most deprived) | 243 | 1019 | 1262
    2 | 749 | 2973 | 3722
    3 | 1172 | 4623 | 5795
    4 | 1193 | 4811 | 6004
    5 (least deprived) | 209 | 847 | 1056
    Missing | 332 | 1298 | 1630

OUTCOME MEASURES:

1. Primary Outcome: Stream 1: Percentage of Participants Who Developed Any Mental Health Condition
Description: Cumulative incidence (percentage of participants in each arm who developed any mental health condition) was calculated using Kaplan-Meier analysis
Time Frame: 5 years
Population: Participants with a pre-existing diagnosis of mental health were excluded
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IBD Cases | Matched Controls
Number analyzed (Participants) | 3423 | 12256
percentage of participants | 12.0 [10.5 to 13.4] | 9.4 [8.7 to 10.1]

2. Primary Outcome: Stream 1: Relative Risk of Any Mental Health Condition
Description: Calculated using Cox proportional hazards models using matched controls as the reference group. Adjusted for age, sex, socioeconomic status, ethnicity, and other common chronic childhood conditions.
Time Frame: Retrospective data assessed from 2010-2020, up to 10 years
Population: Participants with a pre-existing diagnosis of mental health were excluded
Measure: Count of Participants; unit: Participants
Groups:
- Matched Controls (Reference Group): People without a diagnosis in their electronic medical record (ERM) of Inflammatory Bowel Disease, matched on age group, sex, ethnicity (consistent with UK census categories: White, Asian, Black, Mixed, Other), index of multiple deprivation based on postcode, and by practice where numbers allow.
  No specific intervention: Observational analysis of usual care only.
Arm/Group | IBD Cases | Matched Controls (Reference Group)
Number analyzed (Participants) | 3423 | 12256
Participants | 299 | 811
Statistical Analysis 1: Comparison: Matched Controls (Reference Group); Test type: Other; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [1.12 to 1.46] — HR was calculated using a Cox Proportional Hazard model adjusted for age,sex,socioeconomic status, ethnicity and common childhood conditions. Reflects a comparison of the incidence rates between participants diagnosed with IBD and those without IBD

3. Primary Outcome: Stream 2: Relative Risk of Bowel Symptoms (Quality of Life Indicator)
Description: Bowel symptoms consist of abdominal pain, bloating, discomfort and diarrhoea. Relative risk in participants with mental health conditions compared with those without mental health (MH) conditions. Calculated using negative binomial regression.
Time Frame: 5 years of follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- IBD Cases Without Mental Health Condition (Reference Group): A subset of the IBD cases comprising of those participants with the absence of a mental health condition at the same date as their IBD diagnosis. Mental health defined by the diagnosis of any of depression (recurrent depressive disorder or depressive episode), non-phobia-related anxiety disorder (AD), eating disorders, body image disorder, attention-deficit disorder, behavioural disorders, adjustment disorder, acute stress disorder, schizophrenia, bipolar disorder or post-traumatic stress disorder
  No specific intervention: Observational analysis of usual care only.
Arm/Group | IBD Cases With Mental Health Condition | IBD Cases Without Mental Health Condition (Reference Group)
Number analyzed (Participants) | 295 | 1648
Participants | 148 | 473
Statistical Analysis 1: Comparison: IBD Cases Without Mental Health Condition (Reference Group); Test type: Other; Risk Ratio (RR) = 1.82, 95% CI 2-sided [1.33 to 2.52] — RR calculated using negative binomial model adjusted for age,sex,socioeconomic status,ethnicity,IBD type and comorbidities.Reflects a comparison of the incidence rate ratio between IBD participants diagnosed with and without mental health conditions

4. Primary Outcome: Stream 2: Relative Risk of Sleep Disturbance (Quality of Life Indicator)
Description: Relative risk in participants with mental health conditions compared with those without MH conditions. Calculated using Cox regression.
Time Frame: 5 years of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | IBD Cases With Mental Health Condition | IBD Cases Without Mental Health Condition (Reference Group)
Number analyzed (Participants) | 295 | 1648
Participants | 26 | 83
Statistical Analysis 1: Comparison: IBD Cases Without Mental Health Condition (Reference Group); Test type: Other; Hazard Ratio (HR) = 1.63, 95% CI 2-sided [1.02 to 2.62] — HR calculated using Cox regression models adjusted for age,sex,socioeconomic status,ethnicity,IBD type and comorbidities.Reflects a comparison of the incidence rate ratio between IBD participants diagnosed with and without mental health conditions

5. Primary Outcome: Stream 2: Relative Risk of Low Mood (Emotional Function)
Description: Relative risk in participants with mental health conditions compared with those without MH conditions. Calculated using negative binomial regression.
Time Frame: 5 years of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | IBD Cases With Mental Health Condition | IBD Cases Without Mental Health Condition (Reference Group)
Number analyzed (Participants) | 295 | 1648
Participants | 63 | 119
Statistical Analysis 1: Comparison: IBD Cases Without Mental Health Condition (Reference Group); Test type: Other; Risk Ratio (RR) = 2.78, 95% CI 2-sided [1.76 to 4.43] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Stream 1: Lifetime Risk of Developing a Mental Health Condition
Description: Probability of developing a mental health condition by age 25 years.Estimated using modified Cox regression models
Time Frame: Retrospective data assessed from 2010-2020, up to 10 years
Measure: Number; unit: percentage of participants analyzed
Arm/Group | IBD Cases | Matched Controls
Number analyzed (Participants) | 3898 | 15571
percentage of participants analyzed | 31.1 | 25.1

7. Secondary Outcome: Stream 2: Relative Risk of Increased Primary Care Utilisation
Description: Relative risk of increased primary care visits in participants with mental health conditions compared with those without MH conditions. Calculated using negative binomial regression.
Time Frame: 5 years of follow-up.
Measure: Number; unit: Count of prinary care interactions
Arm/Group | IBD Cases With Mental Health Condition | IBD Cases Without Mental Health Condition (Reference Group)
Number analyzed (Participants) | 295 | 1648
Count of prinary care interactions | 12881 | 58153
Statistical Analysis 1: Comparison: IBD Cases Without Mental Health Condition (Reference Group); Test type: Other; Risk Ratio (RR) = 1.33, 95% CI 2-sided [1.12 to 1.58] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Stream 2: Relative Risk of Increased Hospital Admissions
Description: Relative risk of increased hospital admissions in participants with mental health conditions compared with those without MH conditions. Calculated using negative binomial regression.
Time Frame: 5 years of follow-up.
Measure: Number; unit: Count of general hospital admissions
Arm/Group | IBD Cases With Mental Health Condition | IBD Cases Without Mental Health Condition (Reference Group)
Number analyzed (Participants) | 295 | 1648
Count of general hospital admissions | 339 | 1295
Statistical Analysis 1: Comparison: IBD Cases Without Mental Health Condition (Reference Group); Test type: Other; Risk Ratio (RR) = 1.87, 95% CI 2-sided [1.29 to 2.75] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Description: deaths, serious adverse events, and nonserious adverse events were not assessed for study participants
Groups:
- People Diagnosed With Inflammatory Bowel Disease and Presence of a Mental Health Condition: Children, adolescents and young adults (aged 5- 25 years) diagnosed with Inflammatory Bowel Disease (IBD); comprising of Ulcerative Colitis, Crohn's Disease and Unclassified IBD and presence of a diagnosis of a mental health condition.
  Mental health condition comprises any of depression (recurrent depressive disorder or depressive episode), non-phobia-related anxiety disorder (AD), eating disorders, body image disorder, attention-deficit disorder, behavioural disorders, adjustment disorder, acute stress disorder, schizophrenia, bipolar disorder or post-traumatic stress disorder.
- People Diagnosed With Inflammatory Bowel Disease and Absence of a Mental Health Condition: Children, adolescents and young adults (aged 5- 25 years) diagnosed with Inflammatory Bowel Disease (IBD); comprising of Ulcerative Colitis, Crohn's Disease and Unclassified IBD and absence of a diagnosis of a mental health condition.
  Mental health condition comprises any of depression (recurrent depressive disorder or depressive episode), non-phobia-related anxiety disorder (AD), eating disorders, body image disorder, attention-deficit disorder, behavioural disorders, adjustment disorder, acute stress disorder, schizophrenia, bipolar disorder or post-traumatic stress disorder.
Arm/Group | People Diagnosed With Inflammatory Bowel Disease and Presence of a Mental Health Condition | People Diagnosed With Inflammatory Bowel Disease and Absence of a Mental Health Condition
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT05206734/Prot_SAP_001.pdf